CLINICAL TRIAL: NCT01562392
Title: Effects of 5 w Daily Intake of Berries and Vegetables on Cardiometabolic Risk Markers and Cognitive Functions
Brief Title: Effects of Berries and Vegetables on Cardiometabolic Risk Markers and Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Anne Nilsson, PhD, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Dnr 2010/457,2011/510
Record Dates: First submitted 2012-03-15; First posted 2012-03-23 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Metabolic Syndrome; Inflammation; Aging; Fermentation
Keywords: dietary prevention; cognitive performance; metabolic syndrome; colonic fermentation; sub clinical inflammation; cognition and metabolism
MeSH Terms: conditions — Metabolic Syndrome; Inflammation | interventions — Fruit; Vegetables; Control Groups

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- berries and vegetables (Experimental): subjects include specific berries and vegetables in the diet
  Interventions: Dietary Supplement: berries and vegetables
- control product (Placebo Comparator): Control product with equivalent amounts of carbohydrates but without vegetables and berries.
  Interventions: Dietary Supplement: control product

INTERVENTIONS:
Dietary Supplement: berries and vegetables — Daily (5 w) supplementation with specific vegetables and berries
  Arms: berries and vegetables
Dietary Supplement: control product — Supplementation (daily,5 w) with a control product without berries and vegetables.
  Arms: control product

SUMMARY:
The purpose of the study is to study the potential anti-inflammatory- and metabolic effects of polyphenols and dietary fibres in a product based on a mixture of several Swedish berries and vegetables that is known to have high amounts of polyphenols and other anit-oxidants. In addition the purpose is to investigate the effects on cognitive functions of the berry product.

DETAILED DESCRIPTION:
The metabolic syndrome (MetS) includes a cluster of dysfunctions that identifies subjects at risk of developing type-2 diabetes and cardiovascular disease (CVD). A key feature appears to be chronic increased inflammation and activation of the innate system. Consequently, increased low-grade inflammation has been connected to adverse effects on insulin sensitivity, glucose- and lipid metabolism, and blood pressure, and circulating markers of inflammation such as IL-6. A growing body of evidence also link low-grade inflammation to poorer cognitive functioning. Type 2 diabetes, MetS, and glucose intolerance are increasingly being associated with impaired cognition.

Dietary patterns which promote sub-clinical inflammation are increasingly being considered predictive of future risk of CVD and type-2 diabetes. There is a growing insight regarding the role of the colonic micro flora in metabolic regulation and development of low-grade inflammation and obesity. The metabolic cross talk between the colon and peripheral tissues, especially adipose tissue, has been suggested to be regulated through colonic fermentation of indigestible carbohydrates e.g. dietary fibres (DF) and resistant starch. In addition, epidemiological data shows that a high consumption of vegetables and fruits is associated with a lowered risk of cancer and cardiovascular disease, which may be due to the high concentrations of polyphenols or other anti-oxidants that are found in such foods. In addition vegetables and berries are rich in dietary fibres with the potential to beneficially modulate the gut micro flora which may have implication on metabolic risk factors.

In the presently described project it is hypothesized that 5 w daily consumption of a food product containing berries and vegetables can improve metabolic risk variables and cognitive functions. The purpose is therefore to study the potential anti-inflammatory- and metabolic effects, and prebiotic properties, of a food product based on a mixture of several Swedish berries and vegetables that is known to be rich in dietary fibres, polyphenols and other anti-oxidants. In addition the purpose is to investigate the effects on cognitive functions of the food product.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* fasting plasma glucose >6.1
* known cognitive decline
* other medications than for treatment of hypertension or hypothyroidism known gastro- intestinal problems

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Working memory test | 5 week after intervention with test- and control product, respectively
  Cognitive tests (i.e. working memory) will be executed repeatedly in the morning the day after completing the 5 w (35 days)intervention periods.The tests is executed in the morning after a standardised breakfast. The tests starts 30 min after start of the breakfast and are then performed repeatedly at exact time points after the standardised breakfast.The last cognitive test is executed at 150 min post breakfast.

SECONDARY OUTCOMES:
cardiometabolic risk variables | cardiometabolic risk variables will be measured the day for start of and the morning after the 5 week (35 d) intervention periods.
  Inflammatory markers, blood lipids, glucose, insulin, satiety hormons will be determined at fasting in the morning at the first day and the day after completing 5 w (35 days)intervention periods with test product and control product, respectively.
oxidative stress | will be measured the day for start of and the morning after the 5 week (35 d) intervention periods.
  ox-LDL and MDA will be determined in blood at fasting in the morning at the first day and the day after completing 5 w (35 days)intervention periods with test product and control product, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Nutrition and Food Chemistry, Lund University, Lund, Sweden

REFERENCES:
- [Background] Basu A, Du M, Leyva MJ, Sanchez K, Betts NM, Wu M, Aston CE, Lyons TJ. Blueberries decrease cardiovascular risk factors in obese men and women with metabolic syndrome. J Nutr. 2010 Sep;140(9):1582-7. doi: 10.3945/jn.110.124701. Epub 2010 Jul 21. PMID 20660279
- [Background] Krikorian R, Shidler MD, Nash TA, Kalt W, Vinqvist-Tymchuk MR, Shukitt-Hale B, Joseph JA. Blueberry supplementation improves memory in older adults. J Agric Food Chem. 2010 Apr 14;58(7):3996-4000. doi: 10.1021/jf9029332. PMID 20047325
- [Background] Nilsson AC, Ostman EM, Holst JJ, Bjorck IM. Including indigestible carbohydrates in the evening meal of healthy subjects improves glucose tolerance, lowers inflammatory markers, and increases satiety after a subsequent standardized breakfast. J Nutr. 2008 Apr;138(4):732-9. doi: 10.1093/jn/138.4.732. PMID 18356328
- [Derived] Nilsson A, Salo I, Plaza M, Bjorck I. Effects of a mixed berry beverage on cognitive functions and cardiometabolic risk markers; A randomized cross-over study in healthy older adults. PLoS One. 2017 Nov 15;12(11):e0188173. doi: 10.1371/journal.pone.0188173. eCollection 2017. PMID 29141041